CLINICAL TRIAL: NCT01403974
Title: A Phase I Dose Escalation Trial of Weekly Intravenous Administrations of BI 836845 in Patients With Advanced Solid Cancers With Repeated Administrations in Patients Showing Clinical Benefit
Brief Title: Phase I Trial of BI 836845 for Various Solid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1280.1
Record Dates: First submitted 2011-07-12; First posted 2011-07-27 (Estimated); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — xentuzumab

STUDY DESIGN:
Intervention Model Description: Part 1 was conducted in a sequential manner and Part 2 was conducted in a parallel design.

ARMS (16):
- Part 1: BI 836845 10 mg (Experimental): Patients received 10 milligram (mg) of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 20 mg (Experimental): Patients received 20 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 40 mg (Experimental): Patients received 40 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 60 mg (Experimental): Patients received 60 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 90 mg (Experimental): Patients received 90 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 135 mg (Experimental): Patients received 135 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 200 mg (Experimental): Patients received 200 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- Part 1: BI 836845 300 mg (Experimental): Patients received 300 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 450 mg (Experimental): Patients received 450 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 600 mg (Experimental): Patients received 600 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 800 mg (Experimental): Patients received 800 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 1050 mg (Experimental): Patients received 1050 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 1400 mg (Experimental): Patients received 1400 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 1: BI 836845 1800 mg (Experimental): Patients received 1800 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study.
  Interventions: Drug: BI 836845
- Part 2: Ewing's sarcoma family of tumours (Experimental): Patients with Ewing's sarcoma family of tumours (ESFT) receiving relevant biological dose (RBD) of BI 836845 1000 mg, administered in each course of 21 days by a 1-hour infusion at the start of each week in expansion part of the study.
  Interventions: Drug: BI 836845
- Part 2: Biopsiable tumours (Experimental): Patients with all solid tumour types who had tumours suitable for biopsy receiving relevant biological dose (RBD) of BI 836845 1000 mg, administered in each course of 21 days by a 1-hour infusion at the start of each week in expansion part of the study.
  Interventions: Drug: BI 836845

INTERVENTIONS:
Drug: BI 836845 — Intravenous infusion once every week
  Other Names: Xentuzumab

SUMMARY:
This study is a phase I, open-label, dose escalation trial to determine the maximum tolerated dose (MTD) or the relevant biological dose (RBD) in the absence if a MTD of a new drug BI 836845 which blocks the insulin-like growth factor (IGF) pathway believed to be involved in cancer growth. BI 836845 will be administered for the very first time into cancer patients.

The study will also look at the overall safety of the drug, and examine the drug levels in the body at specific timepoints during the trial (pharmacokinetic profile); the effect the drug may have on tumours will also be examined (pharmacodynamics).

ELIGIBILITY:
Inclusion criteria:

1. Patients with histologically or cytologically confirmed diagnosis of advanced, non resectable and / or metastatic solid cancer, who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment.
2. Patients should have evaluable disease, or at least one measurable lesion according to RECIST criteria version 1.1.
3. Age 18 years or older.
4. Life expectancy of at least 3 months in the opinion of the investigator.
5. Written informed consent that is consistent with ICH-GCP guidelines and local legislation.
6. Eastern Cooperative Oncology Group (ECOG) performance score 0, 1 or 2.
7. Patients must have recovered from any previous surgery and have had no major surgery within the last 28 days prior to start of trial medication in the opinion of the investigator.
8. Cardiac left ventricular function with resting ejection fraction > 50% as determined by ECHO or MUGA.
9. Absolute neutrophil count = 1,500/µL.
10. Platelets =100,000/µL.
11. Total bilirubin = 1.5x institution ULN.
12. AST and ALT = 2.5x institution ULN (in case of hepatic primary cancer or known liver metastases: AST and ALT = 5x ULN).
13. Creatinine =1.5 x institution ULN.
14. Haemoglobin = 9g/dL.
15. Haemoglobin A1c less than 8% and fasting plasma glucose =160 mg/dL (=8.9 mmol/L).
16. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) for the duration of trial participation. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days of trial enrolment.
17. Child-Pugh score 5 or 6. (this criterion is limited to HCC patients in Part II only).
18. Patients eligible to undergo tumor biopsy should have normal coagulation parameters (INR and PTT within normal range). (this criterion is limited to patients in Part II only)

Exclusion criteria:

1. Active infectious disease considered by the investigator to be incompatible with the protocol.
2. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol.
3. History of thrombosis (except tumor invading great vessel) within 1 year of study or if concurrent anticoagulation required, except low-dose warfarin (up to 1 mg/day).
4. Patients not recovered from any therapy-related toxicities from previous chemo-, hormone-, immuno-, molecular targeted, or radiotherapies to at least CTCAE = Grade 1. Prior chemotherapy is allowed if completed at least 4 weeks prior to first trial treatment (6 weeks for mitomycin C or nitrosoureas) and the patient has recovered from the acute toxicities of that therapy.
5. Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least 4 weeks before starting trial medication, no history of cerebral oedema or bleeding in the past 4 weeks before starting trial medication and must be on a stable or reducing dose of dexamethasone. Anti-epileptic therapy will be allowed if the patient is stable on antiepileptic treatment for 4 weeks, or more, without adjustments before starting trial medication.
6. Patients who have been treated with any of the following within 4 weeks of starting trial medication: chemotherapy, immunotherapy, radiotherapy, molecular-targeted therapy, biological therapies (including trastuzumab), hormone therapy for breast cancer within 2 weeks of starting trial medication (excluding LHRH agonists in prostate cancer, or bisphosphonates), or treatment with other investigational drugs.
7. Use of any investigational drug within 4 weeks before start of trial medication or concomitantly with this trial.
8. Patients unable to comply with the protocol.
9. Active alcohol abuse or active drug abuse (at the discretion of the investigator).
10. Patients with unstable arrhythmias or unstable angina or severe obstructive pulmonary disease within the last year.
11. For patients entering Part II of the study, prior use of any IGF inhibitor.
12. Pregnancy or breast feeding.
13. Other malignancy requiring active therapy.
14. Patients with a history of diabetes mellitus.
15. For patients that are to undergo tumor biopsy, a history of a hereditary bleeding disorder or clinically relevant major bleeding event in the past 6 months as judged by the investigator (this criterion is limited to patients in Part II only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-07-19 (Actual); Primary Completion 2015-07-08 (Actual); Study Completion 2015-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/ms

REFERENCES:
- [Derived] de Bono J, Lin CC, Chen LT, Corral J, Michalarea V, Rihawi K, Ong M, Lee JH, Hsu CH, Yang JC, Shiah HS, Yen CJ, Anthoney A, Jove M, Buschke S, Fuertig R, Schmid U, Goeldner RG, Strelkowa N, Huang DC, Bogenrieder T, Twelves C, Cheng AL. Two first-in-human studies of xentuzumab, a humanised insulin-like growth factor (IGF)-neutralising antibody, in patients with advanced solid tumours. Br J Cancer. 2020 Apr;122(9):1324-1332. doi: 10.1038/s41416-020-0774-1. Epub 2020 Mar 12. PMID 32161368
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1: dose escalation in patients with advanced solid tumours to determine maximum tolerated dose (MTD) or relevant biological dose (RBD); Part 2: expansion part at the RBD in patients with selected tumour types (Cohort 1- Ewing's sarcoma family of tumours; Cohort 2 - biopsiable solid tumours) in order to investigate safety and pharmacokinetics.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were to be entered to trial drug if any of the specific entry criteria was violated.
Period: Overall Study
Arm/Group | Part 1: BI 836845 10 mg | Part 1: BI 836845 20 mg | Part 1: BI 836845 40 mg | Part 1: BI 836845 60 mg | Part 1: BI 836845 90 mg | Part 1: BI 836845 135 mg | Part 1: BI 836845 200 mg | Part 1: BI 836845 300 mg | Part 1: BI 836845 450 mg | Part 1: BI 836845 600 mg | Part 1: BI 836845 800 mg | Part 1: BI 836845 1050 mg | Part 1: BI 836845 1400 mg | Part 1: BI 836845 1800 mg | Part 2: Ewing's Sarcoma Family of Tumours | Part 2: Biopsiable Tumours
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 1 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 1 | 12
Not completed — Progressive disease according to RECIST | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 6 | 2 | 3 | 2 | 2 | 3 | 1 | 8
Not completed — Dose limiting toxicity (DLT) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Refused to continue study medication | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other than specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: All enrolled patients who gave informed consent and who were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: BI 836845 10 mg | Part 1: BI 836845 20 mg | Part 1: BI 836845 40 mg | Part 1: BI 836845 60 mg | Part 1: BI 836845 90 mg | Part 1: BI 836845 135 mg | Part 1: BI 836845 200 mg | Part 1: BI 836845 300 mg | Part 1: BI 836845 450 mg | Part 1: BI 836845 600 mg | Part 1: BI 836845 800 mg | Part 1: BI 836845 1050 mg | Part 1: BI 836845 1400 mg | Part 1: BI 836845 1800 mg | Part 2: Ewing's Sarcoma Family of Tumours | Part 2: Biopsiable Tumours | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 1 | 12 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 6 | 3 | 4 | 3 | 2 | 3 | 1 | 8 | 50
  >=65 years | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3 | 1 | 2 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 9 | 23
  Male | 2 | 2 | 2 | 0 | 2 | 1 | 2 | 3 | 6 | 2 | 4 | 2 | 3 | 3 | 1 | 3 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 1 | 12 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indian subcontinent Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Southeast Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Japanese | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Korean | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Taiwanese or Chinese | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 1 | 12 | 61
  Asian - other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Maximum Tolerated Dose (MTD) of BI 836845 During the First Treatment Course of the Dose Escalation Phase.
Description: In the absence of MTD, the relevant biological dose (RBD) of BI 836845 during the first treatment course of the dose escalation phase was reported. The MTD was defined as the highest dose level of BI 836845 at which no more than 1 out of 6 patients experienced a drug related dose limiting toxicity (DLT) during the first course of treatment. Starting dose of 10 milligrams (mg) BI 836845, administered thrice every 3 weeks. Dose levels evaluated were: 10 mg, 20 mg, 40 mg, 60 mg, 90 mg, 135 mg, 200 mg, 300 mg, 450 mg, 600 mg, 800 mg, 1050 mg, 1400 mg and 1800 mg.
  The BI 836845 dose which could achieve a plateau in total Insulin-like growth factor 1 (IGF-1) plasma concentrations was considered the RBD.
Time Frame: During the first course of treatment, up to 21 days
Population: Treated set (TS) restricted to the part 1 (dose escalation) of the trial: All enrolled patients who gave informed consent and who were documented to have taken at least one dose of investigational treatment in the dose escalation part of the trial.
Measure: Number; unit: milligram (mg)
Groups:
- Part 1: BI 836845: BI 836845 administered intravenously once every three weeks in patients with advanced solid tumours during dose escalation part of the study
Arm/Group | Part 1: BI 836845
Number analyzed (Participants) | 48
milligram (mg) | 1000

2. Primary Outcome: Part 1: Number of Patients With Dose Limiting Toxicities (DLTs) During the Maximum Tolerated Dose (MTD) Evaluation Period
Description: Number of participants with DLTs occurring during the first treatment course of the dose escalation part. DLT was defined as drug-related adverse events meeting the criteria summarized below:
  * Common terminology criteria for adverse events (CTCAE) grade 4 neutropenia for ≥ 7 days (d)
  * Febrile neutropenia with single temperature of > 38.3°C/ ≥ 38°C more than 1 hour (h)
  * Documented infection with high neutrophile count
  * CTCAE grade 4 thrombocytopenia/CTCAE grade 3 thrombocytopenia associated with bleeding requiring transfusion
  * AST (Aspartate Amino Transferase)/ALT (Alanine Amino Transferase) > 5x normal
  * CTCAE grade 3/4 non-hematologic toxicity
  * CTCAE grade ≥2 infusion reaction
  * CTCAE grade ≥2 nausea and/or vomiting for ≥7 d
  * CTCAE grade ≥3 skin toxicity
  * CTCAE grade ≥3 hyperglycemia
  * Any electrolyte grade 3 AE
  * No recovery from non-DLT CTCAE grade >2
  * Sustained fatigue/asthenia grade 3 for longer than 96 h
  * Other event qualified as DLT by the investigator
Time Frame: During the first course of treatment, up to 21 days
Population: TS restricted to the part 1 (dose escalation) of the trial: All enrolled patients who gave informed consent and who were documented to have taken at least one dose of investigational treatment in the dose escalation part of the trial. Three patients (two patients at the 450 mg and one patient at 800 mg) were replaced thus not included in the analysis of primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BI 836845 10 mg | Part 1: BI 836845 20 mg | Part 1: BI 836845 40 mg | Part 1: BI 836845 60 mg | Part 1: BI 836845 90 mg | Part 1: BI 836845 135 mg | Part 1: BI 836845 200 mg | Part 1: BI 836845 300 mg | Part 1: BI 836845 450 mg | Part 1: BI 836845 600 mg | Part 1: BI 836845 800 mg | Part 1: BI 836845 1050 mg | Part 1: BI 836845 1400 mg | Part 1: BI 836845 1800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Objective Tumour Response Based on Response Evaluation Criteria In Solid Tumours (RECIST) Version 1.1
Description: Number of patients with the objective response (OR). Objective response was defined as best overall response of complete response (CR) or partial response (PR) (with no confirmation required) based on Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1. CR was defined by the disappearance of all target lesions and PR was defined by a decrease of at least 30% in the sum of the diameter of target lesions taking the baseline sum diameters as reference. The best overall response was recorded since first administration of the trial medication and until the earliest of disease progression, death, last adequate tumor assessment or the start of subsequent anti-cancer therapy.
Time Frame: First treatment administration until the earliest of disease progression, death, last adequate tumor assessment or the start of subsequent anti-cancer therapy. Up to 72 weeks.
Population: Treated set (TS): All enrolled patients who gave informed consent and who were documented to have taken at least one dose of investigational treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BI 836845 10 mg | Part 1: BI 836845 20 mg | Part 1: BI 836845 40 mg | Part 1: BI 836845 60 mg | Part 1: BI 836845 90 mg | Part 1: BI 836845 135 mg | Part 1: BI 836845 200 mg | Part 1: BI 836845 300 mg | Part 1: BI 836845 450 mg | Part 1: BI 836845 600 mg | Part 1: BI 836845 800 mg | Part 1: BI 836845 1050 mg | Part 1: BI 836845 1400 mg | Part 1: BI 836845 1800 mg | Part 2: Ewing's Sarcoma Family of Tumours | Part 2: Biopsiable Tumours
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 1 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

4. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response (days), defined as time from first objective response to the time to progression or death and was only calculated for patients with an objective response (with no confirmation required).
Time Frame: as for outcome 3
Population: Treated set (TS): All enrolled patients who gave informed consent and who were documented to have taken at least one dose of investigational treatment. Only two subjects experienced event or were eligible for censoring.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: BI 836845 10 mg | Part 1: BI 836845 20 mg | Part 1: BI 836845 40 mg | Part 1: BI 836845 60 mg | Part 1: BI 836845 90 mg | Part 1: BI 836845 135 mg | Part 1: BI 836845 200 mg | Part 1: BI 836845 300 mg | Part 1: BI 836845 450 mg | Part 1: BI 836845 600 mg | Part 1: BI 836845 800 mg | Part 1: BI 836845 1050 mg | Part 1: BI 836845 1400 mg | Part 1: BI 836845 1800 mg | Part 2: Ewing's Sarcoma Family of Tumours | Part 2: Biopsiable Tumours
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
days |  |  |  |  |  |  |  |  |  |  | 145 [NA to NA] — Only one subject reported OR in this dose group, hence actual duration is presented without confidence interval. | 213 [NA to NA] — Only one subject reported OR in this dose group, hence actual duration is presented without confidence interval. |  |  |  |

5. Secondary Outcome: Best Overall Response Based on Response Evaluation Criteria In Solid Tumours (RECIST) Criteria Version 1.1
Description: Number of patients with best overall response. Best overall response represented the best response (complete response - CR, partial response - PR, stable disease -SD, progressive disease - PD) a patient had during their time in the study from first administration of trial medication until the earliest date of progression, or the last evaluable assessment in the absence of progression or the start of subsequent anti-cancer therapy. CR was defined by the disappearance of all target lesions and PR was defined by a decrease of at least 30% in the sum of the diameter of target lesions taking the baseline sum diameters as reference. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: First treatment administration until disease progression or last evaluable assessment in absence of progression; Up to 72 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Part1: BI 836845 10 mg: Patients received 10 milligram (mg) of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
Arm/Group | Part1: BI 836845 10 mg | Part 1: BI 836845 20 mg | Part 1: BI 836845 40 mg | Part 1: BI 836845 60 mg | Part 1: BI 836845 90 mg | Part 1: BI 836845 135 mg | Part 1: BI 836845 200 mg | Part 1: BI 836845 300 mg | Part 1: BI 836845 450 mg | Part 1: BI 836845 600 mg | Part 1: BI 836845 800 mg | Part 1: BI 836845 1050 mg | Part 1: BI 836845 1400 mg | Part 1: BI 836845 1800 mg | Part 2: Ewing's Sarcoma Family of Tumours | Part 2: Biopsiable Tumours
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 1 | 12
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  SD | 2 | 1 | 2 | 2 | 2 | 0 | 2 | 1 | 3 | 3 | 2 | 0 | 1 | 1 | 1 | 7
  SD≥24 weeks | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  PD | 1 | 2 | 0 | 1 | 1 | 2 | 1 | 2 | 3 | 0 | 1 | 2 | 2 | 2 | 0 | 3
  Not evaluable | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2

6. Secondary Outcome: Disease Control
Description: Number of patients with Disease control. Disease control was defined as best overall response of CR, PR or SD >24 week, with no confirmation required.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BI 836845 10 mg | Part 1: BI 836845 20 mg | Part 1: BI 836845 40 mg | Part 1: BI 836845 60 mg | Part 1: BI 836845 90 mg | Part 1: BI 836845 135 mg | Part 1: BI 836845 200 mg | Part 1: BI 836845 300 mg | Part 1: BI 836845 450 mg | Part 1: BI 836845 600 mg | Part 1: BI 836845 800 mg | Part 1: BI 836845 1050 mg | Part 1: BI 836845 1400 mg | Part 1: BI 836845 1800 mg | Part 2: Ewing's Sarcoma Family of Tumours | Part 2: Biopsiable Tumours
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 1 | 12
Participants | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3

7. Secondary Outcome: Part 2 - Biopsiable Tumours: Progression-free Survival (PFS)
Description: PFS was evaluated only for cohort 2 (Biopsiable tumors) in expansion phase of the study. PFS was defined as the time from first treatment administration until tumour progression according to RECIST 1.1 or death from any cause, whichever occurred earlier. Median duration along with 95% confidence interval is based on Kaplan-Meier method.
Time Frame: First treatment administration until tumour progression or death. Up to 72 weeks
Population: TS restricted to the part 2 - biopsiable tumours cohort (dose expansion) of the trial: All enrolled patients who gave informed consent and who were documented to have taken at least one dose of investigational treatment in the biopsiable tumours cohort of the dose escalation part of the trial.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 2: Biopsiable Tumours
Number analyzed (Participants) | 12
days | 118.0 [18.0 to 504.0]

8. Secondary Outcome: Maximum Measured Concentration of the BI 836845 in Plasma (Cmax)
Description: Maximum measured concentration of the BI 836845 in plasma (Cmax). Geometric mean (gMean) and Geometric coefficient of variation (gCV) is presented for each course. As defined in the CTP, PK data is presented by BI 836845 dose level and was not collected for Course 4 part 2.
  For Course 1 of part 1 and part 2, Course 2 part 1 and part 2, Course 3 part 2, Course 4 part 1 the following timeframe applies : At 0.083 hour before and 0.5, 1, 2, 4, 7, 24, 72*, 168, 169, 336 and 337 hours after infusion. * applies only to part 1 administration courses. In Course 3 of part 1 the following timeframe applies: At 0.083 hour before and 0.5, 1, 168, 169, 336 and 337 hours after infusion.
Time Frame: Up to 337 hours. Detailed timeframe is in the description.
Population: Pharmacokinetic (PK) set: All patients in the treated set who were documented to have received at least one dose of BI 836845 and who had at least one valid PK parameter concentration available. Participants with no available blood samples were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/ml)
Groups:
- Part 2: Expansion Cohort: Patients receiving relevant biological dose (RBD) of BI 836845 1000 mg, administered in each course of 21 days by a 1-hour infusion at the start of each week in expansion part of the study
Arm/Group | Part 1: BI 836845 10 mg | Part 1: BI 836845 20 mg | Part 1: BI 836845 40 mg | Part 1: BI 836845 60 mg | Part 1: BI 836845 90 mg | Part 1: BI 836845 135 mg | Part 1: BI 836845 200 mg | Part 1: BI 836845 300 mg | Part 1: BI 836845 450 mg | Part 1: BI 836845 600 mg | Part 1: BI 836845 800 mg | Part 1: BI 836845 1050 mg | Part 1: BI 836845 1400 mg | Part 1: BI 836845 1800 mg | Part 2: Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 13
microgram per milliliter (µg/ml)
  Course 1 | 2.87 (23.8) | 6.53 (14.9) | 13.8 (26.6) | 22.2 (3.78) | 28.2 (28.7) | 36.6 (20.6) | 70.8 (26.7) | 81.9 (42.2) | 151 (16.7) | 199 (10.8) | 200 (38.1) | 270 (38.9) | 415 (13.0) | 503 (13.4) | 386 (30.7)
  Course 2: number analyzed (Participants) | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 3 | 9
  Course 2 | 3.34 (31.9) | 7.92 (24.8) | 22.4 (23.9) | 26.9 (17.1) | 36.6 (19.4) | 55.2 (29.8) | 99.2 (28.5) | 100 (21.8) | 193 (18.0) | 285 (11.7) | 282 (40.3) | 393 (39.1) | 559 (6.46) | 732 (5.57) | 607 (10.4)
  Course 3: number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 8
  Course 3 | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | 616 (24.8)
  Course 4: number analyzed (Participants) | 2 | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 3 | 3 | 2 | 1 | 1 | 1 | 0
  Course 4 | 3.96 (53.9) | 5.27 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 18.8 (1.88) | 28.5 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 39.6 (15.2) |  | 86.8 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. |  | 201 (10.9) | 279 (28.6) | 253 (36.3) | 615 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 612 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 739 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. |

9. Secondary Outcome: Time to Maximum Measured Concentration BI 836845 in Plasma (Tmax)
Description: Time to maximum measured concentration of the BI 836845 in plasma (tmax). As defined in the CTP, PK data is presented by BI 836845 dose level and was not collected for Course 4 part 2.
  For Course 1 of part 1 and part 2, Course 2 part 1 and part 2, Course 3 part 2, Course 4 part 1 the following timeframe applies : At 0.083 hour before and 0.5, 1, 2, 4, 7, 24, 72*, 168, 169, 336 and 337 hours after infusion. * applies only to part 1 administration courses. In Course 3 of part 1 the following timeframe applies: At 0.083 hour before and 0.5, 1, 168, 169, 336 and 337 hours after infusion.
Time Frame: Up to 337 hours. Detailed timeframe is in the description.
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Groups:
- BI 836845 10 mg: Patients received 10 milligram (mg) of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 20 mg: Patients received 20 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 40 mg: Patients received 40 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 60 mg: Patients received 60 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 90 mg: Patients received 90 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 135 mg: Patients received 135 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 200 mg: Patients received 200 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 300 mg: Patients received 300 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 450 mg: Patients received 450 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 600 mg: Patients received 600 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 800 mg: Patients received 800 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 1050 mg: Patients received 1050 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 1400 mg: Patients received 1400 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- BI 836845 1800 mg: Patients received 1800 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1, 8 and 15 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
- Expansion Cohort: Patients receiving relevant biological dose (RBD) of BI 836845 1000 mg, administered in each course of 21 days by a 1-hour infusion at the start of each week in expansion part of the study
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 60 mg | BI 836845 90 mg | BI 836845 135 mg | BI 836845 200 mg | BI 836845 300 mg | BI 836845 450 mg | BI 836845 600 mg | BI 836845 800 mg | BI 836845 1050 mg | BI 836845 1400 mg | BI 836845 1800 mg | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 13
hours
  Course 1 | 2.10 [1.15 to 4.00] | 2.02 [1.75 to 6.38] | 2.03 [2.00 to 2.03] | 1.13 [1.03 to 1.92] | 2.00 [1.80 to 7.00] | 1.05 [1.03 to 1.92] | 2.00 [2.00 to 3.77] | 2.25 [2.07 to 2.28] | 1.18 [1.02 to 7.00] | 2.00 [1.92 to 2.25] | 1.25 [1.07 to 2.00] | 1.17 [1.02 to 4.02] | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 2.00] | 4.00 [1.00 to 7.00]
  Course 2: number analyzed (Participants) | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 3 | 9
  Course 2 | 0.967 [0.967 to 2.03] | 7.00 [0.967 to 24.1] | 1.50 [1.00 to 2.00] | 2.00 [0.983 to 2.00] | 2.15 [1.00 to 4.00] | 2.89 [1.03 to 4.75] | 2.97 [2.00 to 7.00] | 1.45 [1.05 to 2.02] | 1.12 [1.05 to 2.02] | 2.07 [1.12 to 5.95] | 1.83 [1.40 to 2.00] | 4.00 [3.95 to 4.00] | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 24.0]
  Course 3: number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 8
  Course 3 | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | NA [NA to NA] — Not evaluable due to sparse sampling. | 1.50 [0.983 to 7.00]
  Course 4: number analyzed (Participants) | 2 | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 3 | 3 | 2 | 1 | 1 | 1 | 0
  Course 4 | 3.33 [1.75 to 4.90] | 2.23 [NA to NA] — Only one evaluable subject available for this course in this dose group. Provided Median is actual value, range could not be calculated. | 1.54 [1.08 to 2.00] | 1.02 [NA to NA] — Only one evaluable subject available for this course in this dose group. Provided Median is actual value, range could not be calculated. | 3.09 [2.18 to 4.00] |  | 1.22 [NA to NA] — Only one evaluable subject available for this course in this dose group. Provided Median is actual value, range could not be calculated. |  | 2.00 [1.63 to 7.00] | 2.00 [1.17 to 3.97] | 1.00 [1.00 to 1.00] | 4.00 [NA to NA] — Only one evaluable subject available for this course in this dose group. Provided Median is actual value, range could not be calculated. | 2.00 [NA to NA] — Only one evaluable subject available for this course in this dose group. Provided Median is actual value, range could not be calculated. | 2.00 [NA to NA] — Only one evaluable subject available for this course in this dose group. Provided Median is actual value, range could not be calculated. |

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve of BI 836845 From Time 0 to 168 Hours (AUC 0-168)
Description: Area under the plasma concentration-time curve from time 0 to 168 hours (AUC 0-168) of the BI 836845. As defined in the CTP, PK data is presented by BI 836845 dose level and was not collected for Course 4 part 2.
  For Course 1 of part 1 and part 2, Course 2 part 1 and part 2, Course 3 part 2, Course 4 part 1 the following timeframe applies : At 0.083 hour before and 0.5, 1, 2, 4, 7, 24, 72*, 168, 169, 336 and 337 hours after infusion. * applies only to part 1 administration courses. In Course 3 of part 1 the following timeframe applies: At 0.083 hour before and 0.5, 1, 168, 169, 336 and 337 hours after infusion.
  In the arm BI 836845 450 mg, data from 3 participants was available (15800, 20400 and 12700); as these 3 subjects represented less than 2/3 of the participants included in this course and this dose group, no descriptive statistics were presented in the Clinical Trial Report. The gMean and gCV values were calculated post hoc for ClinicalTrials.gov disclosure purpose only.
Time Frame: Up to 337 hours. Detailed timeframe is in the description.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram hour per milliliter (µg*h/mL)
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 60 mg | BI 836845 90 mg | BI 836845 135 mg | BI 836845 200 mg | BI 836845 300 mg | BI 836845 450 mg | BI 836845 600 mg | BI 836845 800 mg | BI 836845 1050 mg | BI 836845 1400 mg | BI 836845 1800 mg | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 13
microgram hour per milliliter (µg*h/mL)
  Course 1: number analyzed (Participants) | 2 | 3 | 2 | 3 | 3 | 3 | 3 | 2 | 7 | 2 | 3 | 2 | 1 | 1 | 10
  Course 1 | 249 (37.2) | 390 (32.9) | 752 (66.3) | 1300 (42.5) | 2250 (16.7) | 3050 (17.7) | 5950 (26.9) | 5680 (23.1) | 10600 (12.6) | 15600 (7.09) | 14500 (45.6) | 31100 (64.9) | 31800 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 36200 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 32200 (27.4)
  Course 2: number analyzed (Participants) | 3 | 3 | 1 | 1 | 2 | 2 | 3 | 2 | 3 | 2 | 3 | 3 | 3 | 2 | 9
  Course 2 | 265 (49.6) | 627 (41.8) | 1950 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 1790 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 3390 (27.7) | 5150 (52.2) | 9490 (11.1) | 9480 (3.39) | 15997 (24.1) | 21400 (13.0) | 22000 (46.3) | 38600 (34.0) | 48300 (21.7) | 67600 (9.57) | 55500 (20.4)
  Course 3: number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7
  Course 3 | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | NA (NA) — Not evaluable due to sparse sampling. | 53700 (25.4)
  Course 4: number analyzed (Participants) | 2 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0
  Course 4 | 309 (132) | 337 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 1780 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 4010 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 3620 (3.91) |  | 10300 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. |  | 14300 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 17900 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 19000 (78.8) | 56600 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 52400 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. | 67400 (NA) — Only one evaluable subject available for this course in this dose group. Provided gMean is actual value, gCV could not be calculated. |

11. Secondary Outcome: Incidence and Intensity of Adverse Events (AEs) According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
Description: Number of patients with adverse events (AEs) according to the grading as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. The intensity of AEs was defined based on:
  * Grade 1 - Mild AE; awareness of sign(s) or symptom(s) which is/are easily tolerated.
  * Grade 2 - Moderate AE; enough discomfort to cause interference with usual activity.
  * Grade 3 - Severe AE; incapacitating or causing inability to work or to perform usual activities.
  * Grade 4 - Life-threatening or disabling AE.
  * Grade 5 - Death related to AE.
Time Frame: First treatment administration until end of treatment plus residual effect period; Up to 74 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BI 836845 10 mg | Part 1: BI 836845 20 mg | Part 1: BI 836845 40 mg | Part 1: BI 836845 60 mg | Part 1: BI 836845 90 mg | Part 1: BI 836845 135 mg | Part 1: BI 836845 200 mg | Part 1: BI 836845 300 mg | Part 1: BI 836845 450 mg | Part 1: BI 836845 600 mg | Part 1: BI 836845 800 mg | Part 1: BI 836845 1050 mg | Part 1: BI 836845 1400 mg | Part 1: BI 836845 1800 mg | Part 2: Ewing's Sarcoma Family of Tumours | Part 2: Biopsiable Tumours
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 4 | 3 | 3 | 3 | 1 | 12
Participants
  Grade 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Grade 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 4 | 2 | 2 | 1 | 0 | 2 | 1 | 6
  Grade 3 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 3
  Grade 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  Grade 5 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: First treatment administration until end of treatment plus residual effect period; Up to 74 weeks.
Description: Treated set (TS): All enrolled patients who gave informed consent and who were documented to have taken at least one dose of investigational treatment.
Arm/Group | Part 1: BI 836845 10 mg | Part 1: BI 836845 20 mg | Part 1: BI 836845 40 mg | Part 1: BI 836845 60 mg | Part 1: BI 836845 90 mg | Part 1: BI 836845 135 mg | Part 1: BI 836845 200 mg | Part 1: BI 836845 300 mg | Part 1: BI 836845 450 mg | Part 1: BI 836845 600 mg | Part 1: BI 836845 800 mg | Part 1: BI 836845 1050 mg | Part 1: BI 836845 1400 mg | Part 1: BI 836845 1800 mg | Part 2: Ewing's Sarcoma Family of Tumours | Part 2: Biopsiable Tumours
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/3 | 1/3 | 1/3 | 1/3 | 1/3 | 1/3 | 3/8 | 1/3 | 2/4 | 0/3 | 1/3 | 2/3 | 0/1 | 4/12
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 8/8 | 3/3 | 3/4 | 3/3 | 2/3 | 3/3 | 1/1 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: BI 836845 10 mg (N=3) | Part 1: BI 836845 20 mg (N=3) | Part 1: BI 836845 40 mg (N=3) | Part 1: BI 836845 60 mg (N=3) | Part 1: BI 836845 90 mg (N=3) | Part 1: BI 836845 135 mg (N=3) | Part 1: BI 836845 200 mg (N=3) | Part 1: BI 836845 300 mg (N=3) | Part 1: BI 836845 450 mg (N=8) | Part 1: BI 836845 600 mg (N=3) | Part 1: BI 836845 800 mg (N=4) | Part 1: BI 836845 1050 mg (N=3) | Part 1: BI 836845 1400 mg (N=3) | Part 1: BI 836845 1800 mg (N=3) | Part 2: Ewing's Sarcoma Family of Tumours (N=1) | Part 2: Biopsiable Tumours (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: BI 836845 10 mg (N=3) | Part 1: BI 836845 20 mg (N=3) | Part 1: BI 836845 40 mg (N=3) | Part 1: BI 836845 60 mg (N=3) | Part 1: BI 836845 90 mg (N=3) | Part 1: BI 836845 135 mg (N=3) | Part 1: BI 836845 200 mg (N=3) | Part 1: BI 836845 300 mg (N=3) | Part 1: BI 836845 450 mg (N=8) | Part 1: BI 836845 600 mg (N=3) | Part 1: BI 836845 800 mg (N=4) | Part 1: BI 836845 1050 mg (N=3) | Part 1: BI 836845 1400 mg (N=3) | Part 1: BI 836845 1800 mg (N=3) | Part 2: Ewing's Sarcoma Family of Tumours (N=1) | Part 2: Biopsiable Tumours (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 4
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 3 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Miosis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurotrophic keratopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary physical examination abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm of orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.